CLINICAL TRIAL: NCT06720272
Title: Effectiveness of an Integrated Program for the Prevention of Rheumatic Heart Disease in Endemic Regions: a Stepped Wedge Cluster Randomized Trial
Brief Title: School-based Program for the Prevention of Rheumatic Heart Disease in Endemic Regions
Acronym: PREVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Pilgrim (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (CIDRZ) (Unknown); National Academy of Medical Sciences, Nepal (Other Government); University of Oxford (Other)
Responsible Party: Sponsor-Investigator, Thomas Pilgrim, MD, MSc, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: PREVENT
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Rheumatic Heart Disease in Children
Keywords: rheumatic heart disease; valvular heart disease; prevention; streptococcal pharyngitis; rheumatic fever
MeSH Terms: conditions — Rheumatic Heart Disease; Heart Valve Diseases; Rheumatic Fever

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School nurse program (Experimental): The experimental intervention consists in a school nurse program providing integrated health care through diagnosis, intervention, and follow-up of group A beta-hemolytic streptococcal pharyngitis, and facilitation of secondary antibiotic prophylaxis for children with rheumatic heart disease.
  Interventions: Other: School nurse program
- Standard of care (No Intervention): No school nurse prorgam.

INTERVENTIONS:
Other: School nurse program — The intervention consists in the introduction of a school-nurse program providing health care through education about rheumatic heart disease, assessment, intervention, and follow-up of group A beta-hemolytic streptococcal pharyngitis, and facilitation of secondary antibiotic prophylaxis for children with rheumatic heart disease.
  Arms: School nurse program

SUMMARY:
The overall objective of the PREVENT trial is to evaluate the effectiveness of an integrated, school-based program for the prevention of rheumatic heart disease (RHD) in regions with an endemic pattern of RHD.

We conduct a stepped wedge cluster randomized trial in randomly selected schools in Nepal and Zambia.

The intervention will be delivered at the level of the school and consists in the introduction of a dedicated school-nurse program providing health care through education about RHD, assessment, intervention, and follow-up of GABHS pharyngitis, and facilitation of secondary antibiotic prophylaxis for children with RHD.

ELIGIBILITY:
Inclusion Criteria:

- Children aged 5-16 years

Exclusion Criteria:

* Children / primary caregivers not providing informed consent to participate
* Children not attending one of the selected schools

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6000 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Rheumatic heart disease | The endpoint will be assessed after a minimum of 1 and a maximum of 3 years after introduction of the school nurse program.
  The primary outcome of the study will be the reduction in prevalence of rheumatic heart disease according to WHF criteria 2023 as assessed by systematic echocardiographic screening.

CONTACTS AND LOCATIONS:
Locations (2):
- National Academy od Medical Sciences, Kathmandu, Nepal
- Centre of Infectious Disease Research, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided